CLINICAL TRIAL: NCT02074410
Title: Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Safety and Efficacy of OMS643762 in Subjects With Huntington's Disease
Brief Title: Safety and Efficacy of OMS643762 in Subjects With Huntington's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision - pending further analysis of available data
Sponsor: Omeros Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OMS824-HTD-002
Record Dates: First submitted 2014-02-21; First posted 2014-02-28 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Huntington's Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- OMS643762 Low Dose without food (Experimental): Orally administering OMS643762 low dose daily without food for 28 days
  Interventions: Drug: OMS643762
- OMS643762 Medium Dose without food (Experimental): Orally administering OMS643762 medium dose daily without food for 28 days
  Interventions: Drug: OMS643762
- OMS643762 Medium Dose with food (Experimental): Orally administering OMS643762 Medium dose daily with food for 28 days
  Interventions: Drug: OMS643762
- Placebo (Placebo Comparator): Orally administering placebo daily for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OMS643762
  Other Names: OMS824
  Arms: OMS643762 Low Dose without food; OMS643762 Medium Dose with food; OMS643762 Medium Dose without food
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety, tolerability and pharmacokinetics of OMS643762 (the study drug) in subjects with Huntington's disease (HD).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily provide informed consent, or have a legally authorized representative (LAR) provide informed consent with subject assent, in accordance with local regulations and governing Institution Review Board (IRB) requirements prior to any procedures or evaluations performed specifically for the sole purpose of the study (other than the Montreal Cognitive Assessment (MoCA) to assess capacity to provide informed consent). Capacity to provide informed consent will be determined by the MoCA and investigator judgment according to the following:

   * Subjects with scores of greater than or equal to 21 on the MoCA and, in the judgment of the investigator, have the capacity to provide valid informed consent, can give consent.
   * Subjects with scores of less than 21 but greater than or equal to 18 on the MoCA and, in the judgment of a mental health professional (independent of the investigator) have the capacity to provide valid informed consent, may give consent.
   * Subjects with scores less 21 but greater than or equal to 18 on the MoCA, who lack the capacity to give valid informed consent, in the judgment of a mental health professional (independent of the investigator), will need an LAR to provide informed consent with assent by the subject.
   * Subjects with scores of less than 18 on the MoCA will have an LAR provide informed consent with assent by the subject.
2. Have a clinical diagnosis of HD, confirmed by either CAG repeat number of greater than or equal to 39 or a positive family history (a first degree relative with a clinical diagnosis of HD) if CAG repeat number is not known.
3. Are age greater than or equal to 18 and less than or equal to 65 years at the screening visit (Visit 1).
4. Have a UHDRS Total Functional Capacity greater than or equal to 7 at Visit 1.
5. If currently taking antipsychotic medication(s), have been on a stable regimen for at least 60 days prior to randomization.
6. Are fluent in English.
7. If female, are either a) not of childbearing potential (i.e., surgically sterilized or post-menopausal for more than 1 year) or b) have a negative pregnancy test and if sexually active must agree to use a medically reliable form of contraception throughout the study. Acceptable methods of contraception include a reliable intrauterine device, hormonal contraception or spermicide in combination with a barrier method.
8. If male, are either a) not of reproductive potential or b) if sexually active must agree to use a medically reliable form of contraception throughout the study. Acceptable methods of birth control include spermicide in combination with a barrier method, or subjects' female partner is willing to use medically acceptable methods of birth control.
9. Have normal clinical laboratory test results and ECG, or results with minor deviations, which are not considered to be clinically significant by the investigator.

Exclusion Criteria:

1. Have a history or presence of significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, or neurological disorders other than HD which, in the opinion of the investigator, increases the risk of the study drug or may confound the interpretation of study measures.
2. Have unstable or severe depression, in the opinion of the investigator.
3. Have alcohol or drug abuse or dependence, as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision.
4. Have received treatment with an investigational drug or device within 60 days prior to Visit 1.
5. Are pregnant or lactating.
6. Have serum alanine transaminase or aspartate transaminase greater than two times upper limit of normal at screening.
7. Have hemoglobin, white blood cell count, absolute neutrophil count, or platelet count outside the normal range at screening.
8. Are an employee of Omeros, an investigator, or study staff member, or their immediate family member.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10-15 (Actual); Study Completion 2014-10-15 (Actual)

PRIMARY OUTCOMES:
Assess the Safety of OMS643762 | 28 days
  Safety as assessed by adverse events
Assess the Safety of OMS643762 | 28 days
  Safety as assessed by vital signs
Assess the Safety of OMS643762 | 28 days
  Safety as assessed by clinical lab-tests
Assess the Safety of OMS643762 | 28 days
  Safety as assessed by ECG
Assess the Safety of OMS643762 | 28 days
  Safety as assessed by Columbia-Suicide Severity Rating Scale (C-SSRS)

SECONDARY OUTCOMES:
Motor function | Pre-dose and day 15 and 28 post-dose
  Change from baseline in the UHDRS - Total Motor Score
Motor function | Pre-dose and day 15 and 28 post-dose
  Change from baseline in the Speeded Tapping Test score
Cognition | Pre-dose and day 28 post-dose
  Change from baseline in the Cognitive Assessment Battery composite score
Behavior | Pre-dose and day 28 of dosing
  Change from baseline in the Problem Behavior Assessment score
Pharmacokinetics profile | Pre-dose, day 15 and 28 of dosing and up to 14 days post-dose
  Maximum plasma concentration of OMS643762 following multiple-dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Steve Whitaker, MD, Study Director — Omeros Corporation
Locations (9):
- United States (9):
  - San Diego, California
  - Englewood, Colorado
  - Gainesville, Florida
  - Tampa, Florida
  - Baltimore, Maryland
  - New York, New York
  - Memphis, Tennessee
  - Houston, Texas
  - Kirkland, Washington